CLINICAL TRIAL: NCT02011867
Title: A New Cochlear Implant Electrode With A "Cork" Type Stopper For Inner Ear Malformations
Brief Title: A New Cochlear Implant Electrode For Inner Ear Malformations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Münir Demir Bajin, MD, Hacettepe University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO-13/315
Record Dates: First submitted 2013-11-30; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Inner Ear Malformations
Keywords: Inner Ear Malformations; Gusher; Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cork Electrode (Experimental): Using Cork Electrode for CSF leak prevention for inner ear malformations.
  Interventions: Device: Cork Electrode

INTERVENTIONS:
Device: Cork Electrode
  Other Names: MedEl Cork Electrode

SUMMARY:
The custom made device was produced by Med-El Company. It has a "cork" like stopper instead of the usual silicon ring to prevent gusher. There are two types of electrodes consisting of different length. Standard one is 25 mm (contact space 1.7 mm) and the short one is 20 mm (contact space 1.3 mm). It was used in 50 patients with different inner ear malformations. Thirteen patients had gusher, and 11 patients oozing during cochleostomy. One patient with initial prototype of the cork electrode had to be revised because of persistent oozing around the electrode. Another patient had slow extrusion of the electrode most probably due to CSF (cerebrospinal fluid) pulsation and had to be revised. Both patients had no more CSF fistula.

CSF fistula in inner ear malformations is a serious situation which may lead to recurrent meningitis. The new cochlear implant electrode with "cork" stopper looks promising in preventing the postoperative CSF leak around the electrode.

DETAILED DESCRIPTION:
Gusher in inner ear malformations is common in patients with incomplete partition type-I, and III. It is also common in less severe form as oozing in incomplete partition type II and large vestibular aqueduct. It is important to prevent CSF escape around the cochlear implant electrode to prevent meningitis.

The custom made device was produced by Med-El Company. It has a "cork" like stopper instead of the usual silicon ring to prevent gusher. There are two types of electrodes consisting of different length. Standard one is 25 mm (contact space 1.7 mm) and the short one is 20 mm (contact space 1.3 mm). It was used in 50 patients with different inner ear malformations.

Thirteen patients had gusher, and 11 patients oozing during cochleostomy. One patient with initial prototype of the cork electrode had to be revised because of persistent oozing around the electrode. Another patient had slow extrusion of the electrode most probably due to CSF pulsation and had to be revised. Both patients had no more CSF fistula.

CSF fistula in inner ear malformations is a serious situation which may lead to recurrent meningitis. The new cochlear implant electrode with "cork" stopper looks promising in preventing the postoperative CSF leak around the electrode.

ELIGIBILITY:
Inclusion Criteria:

* Must have an inner ear malformation
* Must meet the criteria for cochlear implantation

Exclusion Criteria:

* Prior cochlear implantation surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
CSF leak | Up to 1 year
  Occurrence of CSF leak after the surgery.

SECONDARY OUTCOMES:
Meningitis | Up to 1 year
  Having meningitis due to CSF leak or connection to the middle ear after surgery.

OTHER OUTCOMES:
Hearing | Until death
  Improvement in hearing after cochlear implantation.